CLINICAL TRIAL: NCT07248384
Title: The Efface of Ketamine vs. Lidocaine in the Management of Pain After Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: The Efface of Ketamine vs. Lidocaine in the Management of Pain After Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Mustafa Hussain Imam, Mustafa Hussain Imam, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1097-2024-LNH-ERC
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pain, Postoperative
Keywords: Ketamine; Lidocaine; Postoperative Pain; Pain; Laparoscopic Cholecystectomy; Analgesia; Visual Analogue Scale (VAS); Anesthesia; Pain Management
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine Group (Active Comparator): The ketamine dose was calculated as 0.5 mg/kg of body weight, diluted with normal saline to a total volume of 10 mL, and administered intravenously as a stat dose during anesthesia reversal, following the completion of surgery.
  Interventions: Drug: IV ketamine 0.5 mg/kg
- Lidocaine Group (Active Comparator): A total of 3 mL of 2% lidocaine was diluted with 7 mL of normal saline to prepare a 10 mL solution, which was administered intravenously as a stat dose at the time of anesthesia reversal, immediately after completion of surgery.
  Interventions: Drug: IV Lidocain 60 mg/kg

INTERVENTIONS:
Drug: IV ketamine 0.5 mg/kg — Patients in the Ketamine group received intravenous ketamine at a dose of 0.5 mg/kg body weight, diluted with normal saline to a total volume of 10 mL. The prepared solution was administered as a single (stat) intravenous injection at the time of anesthesia reversal, immediately after completion of laparoscopic cholecystectomy. The drug was administered under aseptic precautions by an anesthetist who was blinded to group allocation.
  All patients received standard postoperative care, including intravenous diclofenac sodium 75 mg every 8 hours for baseline analgesia and ondansetron 4 mg IV for nausea prevention. Postoperative pain intensity was recorded at 1, 6, 12, and 24 hours using the Visual Analogue Scale (VAS). Patients reporting significant pain were administered intravenous Kinz 5 mg as rescue analgesia, and the timing of administration was documented.
  Arms: Ketamine Group
Drug: IV Lidocain 60 mg/kg — Patients in the Lidocaine group received 3 mL of 2% lidocaine, diluted with 7 mL of normal saline to prepare a 10 mL solution, which was administered intravenously as a stat dose at the time of anesthesia reversal, immediately after surgery. The intervention was given using the same protocol and blinding method as the Ketamine group to maintain uniformity.
  Similar to Group K, all patients received standard postoperative medications, including IV diclofenac sodium and ondansetron. Pain assessment was performed using the VAS scale at 1, 6, 12, and 24 hours postoperatively. Patients requiring additional pain relief were given IV Kinz 5 mg as rescue analgesia, with the time of each administration noted.
  Arms: Lidocaine Group

SUMMARY:
This prospective interventional study conducted at Liaquat National Hospital and Medical College compared the analgesic efficacy of ketamine and lidocaine in managing postoperative pain after laparoscopic cholecystectomy. Total of 76 ASA I-II patients were randomly assigned into two equal groups (Group K: Ketamine, Group L: Lidocaine) using a sealed-envelope method in a double-blind, placebo-controlled design. Standard anesthesia with propofol, isoflurane, and atracurium was administered, and all patients received postoperative diclofenac sodium and ondansetron. Pain intensity was assessed using the Visual Analogue Scale (VAS) at 1, 6, 12, and 24 hours postoperatively. The study aimed to compare the pain-relieving effects of ketamine and lidocaine, contributing to improved strategies for postoperative pain management following laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Effective postoperative pain management is essential for promoting patient recovery, reducing stress response, and improving overall outcomes following laparoscopic cholecystectomy. This prospective interventional study was conducted at Department of Anesthesiology at Liaquat National Hospital and Medical College to compare the analgesic efficacy of intravenous ketamine and lidocaine in managing postoperative pain among patients undergoing elective laparoscopic cholecystectomy.

A total of 76 ASA grade I and II patients with uncomplicated symptomatic gallstone disease were enrolled after obtaining written informed consent and ethical approval. Using a sealed-envelope randomization method, patients were divided into two equal groups: Group K (n=38) received ketamine, and Group L (n=38) received lidocaine. The study followed a double-blinded, placebo-controlled design to ensure unbiased assessment. Patients with ASA grade III-V, chronic pain, psychiatric illness, pregnancy or lactation, major hepatic, renal, or cardiovascular dysfunction, or a recent history of opioid or NSAID use were excluded.

All participants underwent standard preoperative preparation, including overnight fasting and pre-anesthetic evaluation. General anesthesia was induced with propofol and atracurium and maintained with isoflurane. Standard intraoperative monitoring of pulse rate, blood pressure, ECG, SpO₂, and end-tidal CO₂ was performed. Following surgery, residual neuromuscular blockade was reversed with neostigmine. All patients received intravenous diclofenac sodium every 8 hours for baseline analgesia and ondansetron to prevent postoperative nausea and vomiting.

Pain intensity was assessed using the Visual Analogue Scale (VAS) at 1, 6, 12, and 24 hours postoperatively. Patients who reported pain received intravenous Kinz 5 mg as rescue analgesia, with timing recorded by nursing staff.

This study provided valuable insight into the comparative analgesic effects of ketamine and lidocaine for postoperative pain control following laparoscopic cholecystectomy, emphasizing their potential role in multimodal analgesia protocols to enhance patient comfort and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.

ASA physical status I-II.

Elective laparoscopic cholecystectomy planned under general anesthesia.

Normal baseline renal, hepatic, and coagulation profile.

Able to give informed consent and communicate pain scores.

Negative pregnancy test for women of childbearing age.

Exclusion Criteria:

* ASA III-V patients.

Allergy or hypersensitivity to ketamine, lidocaine, or related drugs.

History of psychiatric illness or substance abuse.

Chronic use of opioids, benzodiazepines, or MAO inhibitors.

Pregnant or breastfeeding women.

Chronic pain disorders or use of analgesics within 7 days pre-op.

Major hepatic, renal, or cardiovascular dysfunction.

History of myopathy or seizure disorders.

Patients with atrioventricular block or on calcium-channel blockers.

Conversion to open cholecystectomy during surgery.

Inability to understand or report pain postoperatively.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Score | Postoperative pain was assessed at the 1st, 6th, 12th, and 24th hours.
  Postoperative pain intensity was assessed using the Visual Analogue Scale (VAS) at 1, 6, 12, and 24 hours after surgery to evaluate and compare the effectiveness and duration of analgesia between the ketamine and lidocaine groups. These time intervals were selected to monitor both the early and late postoperative pain responses during the first 24 hours of recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Hussain Imam, Mbbs, Principal Investigator — Liaquat National Hospital
Locations (1):
- Liaquat National Hospital, Anesthesiology Department, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No